CLINICAL TRIAL: NCT05625893
Title: Proton Beam Radiotherapy Followed by Tecentriq and Avastin for Primary Liver Cancer With Vp2-4 Portal Vein Invasion: PORTAL Study
Brief Title: Proton Beam Radiotherapy Followed by Tecentriq and Avastin for Primary Liver Cancer With Vp2-4 Portal Vein Invasion
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Il Yu, Assistant Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PORTAL
Record Dates: First submitted 2022-09-20; First posted 2022-11-23 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Thrombosis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PBT arm (Experimental)
  Interventions: Radiation: PBT and atezolizumab/bevacizumab

INTERVENTIONS:
Radiation: PBT and atezolizumab/bevacizumab — Atezolizumab 1200 mg and bevacizumab 15 mg/Kg is administered IV infusion every 3 weeks.
  Proton beam therapy 30 - 50 Gy/5 fractions to portal vein tumor thrombosis with or without main primary tumor after 1 week (+/- 7 days) of 2nd cycle of atezolizumab and bevacizumab
  The follow-up phase begins when the decision to discontinue study is made. The follow-up phase is defined as the day after the end of study treatment until the day the subject dies.

SUMMARY:
This study is investigator initiated, single-institution, prospective, phase 2 open-label study to determine the efficacy and safety of combination therapy of atezolizumab/bevacizumab and proton beam therapy to portal vein tumor thrombosis with or without main primary tumor in patients with stage 3 or higher hepatocellular carcinoma (HCC) with Vp2-4 portal vein invasion who had not undergone systemic therapy for HCC. The primary endpoint of this study is progression-free survival and secondary endpoints are overall survival (OS), time to progression (TTP), objective response rate, disease control rate (DCR), and time to local disease progression (LTP).

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCC meeting all of following criteria;

  1. Histologically or radiologically confirmed hepatocellular carcinoma based on the guidelines of the Korean Liver Cancer Association-National Cancer Center 2022
  2. Age >= 20
  3. Vp2-4 portal vein tumor thrombosis diagnosed by dynamic enhanced computed tomography (CT) or maganetic resonance images (MRI) with below finding 1) an intraluminal filling defect adjacent to the primary tumor in Vp2-4 portal vein 2) an enhancement of the filling defect on arterial phase and a washout on portal/delayed phases.
  4. Signed written informed consent
  5. at least one or more measurable intrahepatic viable HCC lesions
  6. Child-Pugh class A within 2 weeks from screening for study registration
  7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1 within 2 weeks from screening for study registration
  8. Life expectancy of at least 16 weeks
  9. adequate bone marrow and liver function within 2 weeks from screening for study registration

     * Hemoglobin ≥ 9.0 g/dL

       * Absolute neutrophil count (ANC) ≥ 1,000/mm3

         * Platelet count ≥ 50,000/μL

           * Total bilirubin < 2.5 mg/dL

             * Serum albumin >2.8 g/dL

               * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × upper limit of normal (ULN)

                 * Prothrombin time in INR ≤ 1.8 × ULN

                   * Serum creatinine ≤ 1.5 mg/dL
  10. Women of childbearing potential and men must agree to use highly efficient contraception since signing of the informed consent form until at least 6 months (women) and 7 months (men) after the last study drug administration
  11. If other selection conditions are satisfied and the exclusion criteria are not met, registration is possible even in case of N1 or M1.
  12. Registration is possible even in the case of hepatic vein tumor infiltration if other selection conditions are satisfied and the exclusion criteria are not met
  13. no limitation according to the size and number of tumors in the liver.

Exclusion Criteria:

Patients with HCC meeting all of following criteria;

1. previous history of systemic treatment for HCC (If systemic treatment for HCC has been performed at least once, it will not be enrolled in this study.) However, registration is permitted if the previous systemic treatment is for adjuvant purposes or treatment for other cancers. Also allowed if previous HCC treatment is local treatment. However, cases with a history of previous upper abdominal radiotherapy (including proton therapy and heavy particle therapy) are excluded.
2. any type of anticancer agent (including investigational) within 2 weeks before enrollment
3. Having active brain metastasis or leptomeningeal metastasis need surgery or steroid therapy
4. Moderate to severe or intractable ascites
5. A history or presence of hepatic encephalopathy
6. Presence of active bacterial infection
7. Untreated active chronic hepatitis B or active hepatitis C
8. History of portal hypertension with bleeding within the past 6 months
9. Prior liver transplant
10. Uncontrolled severe medical comorbidity
11. unhealed wound
12. uncontrolled electrolyte imbalance
13. Non-interruptible therapeutic use of anticoagulants or thrombolytics
14. History of uncontrolled or autoimmune disease, or immunocompromised
15. interstitial lung disease
16. Other malignant disease (a history of treated malignancy -other than HCC- is allowable if the patient's malignancy has been in complete remission, off chemotherapy and without additional surgical intervention, during the preceding two years)
17. Mentally retarded/medically incapable of consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | At 9 month
Incidence of adverse event assessed according to the Common Terminology Criteria for Adverse Events (CTCAE version 5.0) | From date of atezolizumab and bevacizumab initiatton until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months

SECONDARY OUTCOMES:
Overall survival rate | At 12 month
Time-to-progression | At 9 months
Objective response rate | At 3 month
Disease Control rate | At 3 month
Local tumor progression rate | At 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Il Yu, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided